CLINICAL TRIAL: NCT01038362
Title: Effects Of Almonds On Vascular Reactivity And Biomarkers Of Inflammation, Oxidative Stress And Endothelial Function In Patients With Coronary Artery Disease
Brief Title: Effects of Almonds On Endothelial Function In Patients With Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Tufts University (Other)
Responsible Party: Joseph A. Vita, MD, Boston University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: H-27411
Record Dates: First submitted 2009-12-19; First posted 2009-12-23 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Coronary Artery Disease
Keywords: endothelium; almonds; dietary interventions; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Almonds (Active Comparator): National Cholesterol Education Program Step I diet plus almonds for 6 weeks
  Interventions: Other: NCEP Step 1 diet plus Almonds
- No Almonds (Placebo Comparator): National Cholesterol Education Program Step 1 diet without almonds for 6 weeks
  Interventions: Other: No Almonds

INTERVENTIONS:
Other: NCEP Step 1 diet plus Almonds — NCEP Step 1 Diet Plus Almonds 3 oz per day for 6 weeks
  Arms: Almonds
Other: No Almonds — NCEP Step 1 diet without almonds
  Arms: No Almonds

SUMMARY:
The vascular endothelium (inner lining of cells in blood vessels) normally prevents vasospasm and thrombosis by production of a variety of regulatory substances, including nitric oxide. In patients with atherosclerosis, these functions of the endothelium are impaired and these abnormalities may contribute to the development of heart attack and stroke.

Observational studies have shown that frequent nut consumption decreases the risk of cardiovascular disease (CVD), but the mechanisms of benefit have not been fully defined. Recent studies suggest that specific fatty acids and flavonoids in nuts may have favorable effects on cardiovascular disease. In addition, there is growing evidence that these compounds may improve the function of the endothelium.

The present study is designed to test the hypothesis that an almond-enriched diet will improve the function of the endothelium in patients with coronary artery disease. Subjects will be enrolled into a randomized, placebo-controlled, crossover study that will compare a National Cholesterol Education Program Step 1 diet without nuts to a Step 1 diet that has the same number of total calories but includes 3 ounces of almonds daily. Participants will consume each diet for six weeks with a four-week rest period between diets. The order of diets will be randomized (almonds or no almonds). Dietary assessments via food recall questionnaires will be employed at the study entry, end of the four week washout period, and end of the second intervention. If subjects are drifting from the recommendations of the STEP 1 diet, counseling will be given to urge compliance. The primary endpoint will be endothelium-dependent flow- mediated dilation assessed by ultrasound. Secondary study outcomes will include lipid profiles, markers of inflammation and oxidative stress. Enrollment will continue until 40 subjects with complete data are available.

Patients will be enrolled at Boston Medical Center and the Jean Mayer US Department of Agriculture Human Nutrition Research Center at Tufts Medical Center. Dietary interventions will be performed at Tufts Medical Center or by telephone. Ultrasound studies and blood collection will be performed in the principal investigator's research unit at Boston Medical Center.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female subjects.
2. Age range: 21-80 years old.
3. Weight less than 115 kg.
4. Clinically defined coronary artery disease that is clinical stable and compensated with appropriate treatment. Coronary disease (CVD) is defined by the presence of lesions on coronary angiography, history of myocardial infarction, or positive stress test.
5. Willingness to give written informed consent and willingness and ability to understand, to participate to and to comply with the study requirements.

Exclusion Criteria:

1. History of nut allergy.
2. Pregnant or lactating women. Pregnancy will be excluded by urine pregnancy test.
3. Clinical history of other major illness including end-stage cancer, renal failure, hepatic failure, gastrointestinal disorders that may impair absorption, or other conditions that in the opinion of the principal investigator make a clinical study inappropriate.
4. Treatment with an investigational new drug within the last 30 days.
5. History of a psychological illness or condition such as to interfere with the subject's ability to understand the requirements of the study.
6. Unwillingness to comply with the requirements of study including refraining from consumption of nuts and refraining from use of Vitamin E, vitamin C, and beta carotene, lipoic acid, and/or other dietary or herbal supplements during the study.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation | 6 weeks

SECONDARY OUTCOMES:
Blood markers of inflammation, dyslipidemia, and oxidative stress | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Vita, MD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States